CLINICAL TRIAL: NCT04565717
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, 3-Part Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Dose ALN-HSD in Healthy Adult Subjects and Multiple Dose ALN-HSD in Adult Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study of ALN-HSD in Healthy Adult Subjects and Adult Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study ALN-HSD-001 was terminated due to business reasons and changes in the development strategy of the product. No safety issues were found.
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-HSD-001; 2020-000847-29 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Nonalcoholic Steatohepatitis; NASH
Keywords: Hepatobiliary disorders; Non-alcoholic fatty liver disease; NAFLD; Fatty liver; RNAi therapeutic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Digestive System Diseases; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts A&B: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor); Part C: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: ALN-HSD (Experimental): Participants will be administered a single dose of ALN-HSD.
  Interventions: Drug: ALN-HSD
- Part A: Placebo (Placebo Comparator): Participants will be administered a single dose of ALN-HSD-matching placebo.
  Interventions: Drug: Placebo
- Part B: ALN-HSD (Experimental): Participants will be administered multiple doses of ALN-HSD.
  Interventions: Drug: ALN-HSD
- Part B: Placebo (Placebo Comparator): Participants will be administered multiple doses of ALN-HSD-matching placebo.
  Interventions: Drug: Placebo
- Part C: ALN-HSD (Experimental): Participants will be administered multiple doses of ALN-HSD.
  Interventions: Drug: ALN-HSD

INTERVENTIONS:
Drug: ALN-HSD — ALN-HSD will be administered by subcutaneous (SC) injection.
  Arms: Part A: ALN-HSD; Part B: ALN-HSD; Part C: ALN-HSD
Drug: Placebo — Normal saline (0.9% NaCl) matching volume of ALN-HSD doses will be administered SC.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending doses of ALN-HSD in healthy participants (Part A) and multiple doses of ALN-HSD in patients with NASH (Parts B and C).

ELIGIBILITY:
Inclusion Criteria:

* Part A Only

  * Has body mass index (BMI) ≥18 kg/m^2 and ≤28 kg/m^2
  * Has normal 12-lead electrocardiogram (ECG)
* Parts B and C Only:

  * Has BMI ≥18 kg/m^2 and ≤40 kg/m^2
  * Has a diagnosis of NASH documented in the patient's medical history or a clinical suspicion of NASH based on defined study criteria
  * Has screening liver biopsy with NASH activity score (NAS) score of ≥3 per NASH Clinical Research Network (CRN) criteria

Exclusion Criteria:

* Parts A, B and C:

  * Has any clinical safety laboratory result considered clinically significant and unacceptable by the Investigator
  * Has known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
  * Has known history or evidence of drug abuse, within 12 months prior to screening
  * Has evidence of other forms of known chronic liver disease
  * Has recently received an investigational agent
  * Has any uncontrolled or serious disease, medical or surgical condition that my interfere with participation or data interpretation
  * Has excessive alcohol intake for ≥ 3 months during past year
  * Has history of intolerance to SC injection(s)
  * Has international normalized ratio (INR) >1.2
  * Has platelet count <140x10^9/L
* Part A Only

  * Has systolic blood pressure (BP) >140 mmHg and diastolic >90 mmHg;
  * Has used certain prescription drugs within last 14 days prior to screening
  * Has used certain over the counter (OTC) medication within 7 days prior to screening
  * Has estimated glomerular filtration rate (GFR) <90 mL/min/1.73m^2 at screening
* Parts B and C Only

  * Has abnormal ECG
  * Has changes in certain prescription medications defined in the protocol within the specified timeframe prior to screening
  * Has GFR<45ml/min/1.73m^2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Frequency of Adverse Events | Part A: Up to 3.5 months; Part B: up to 12.5 months
Part C: Change from Baseline of Liver Hydroxysteroid 17β Dehydrogenase 13 (HSD17B13) Messenger Ribonucleic Acid (mRNA) | Baseline and Month 6

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Concentration-time Curve (AUC) for ALN-HSD and Potential Metabolites | Day 1 predose and up to 48 hours postdose
Pat A: Maximum Plasma Concentration (Cmax) for ALN-HSD and Potential Metabolites | Day 1 predose and up to 48 hours postdose
Part A: Fraction Excreted in Urine (fe) of ALN-HSD and Potential Metabolites | Day 1 up to 24 hours postdose
Part B: Plasma Concentrations of ALN-HSD and Potential Major Metabolite(s) | Day 1 and Month 3 predose and up to 4 hours postdose
Part B: Change from Baseline of Liver HSD17B13 mRNA | Predose and up to 9 months postdose
  Hepatic HSD17B13 mRNA will be measured by quantitative reverse-transcription polymerase chain reaction using ribonucleic acid (RNA) isolated from liver biopsy.
Part C: Frequency of Adverse Events | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (11):
- United States (5):
  - Clinical Trial Site, Fleming Island, Florida
  - Clinical Trial Site, Marrero, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Hermitage, Tennessee
  - Clinical Trial Site, San Antonio, Texas
- Clinical Trial Site, Brussels, Belgium
- Clinical Trial Site, Sofia, Bulgaria
- Turkey (Türkiye) (2):
  - Clinical Trial Site, Balçova
  - Clinical Trial Site, Izmir
- United Kingdom (2):
  - Clinical Trial Site, Edinburgh
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232